CLINICAL TRIAL: NCT06678386
Title: Alteration of Sweet Taste Perception After 50% Reduction of Sweet Food and Beverage Consumption for 12 Weeks, Compared With Unmodified Diet.
Brief Title: Alteration of Sweet Taste Perception After Reduction of Sweet Food and Beverage Consumption.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 233/2567 (IRB1)
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Health-Related Behavior
Keywords: sweet taste perception; sugar reduction; dietary behavior; dietary modification; sweet intensity
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50% sugar reduction (Experimental): Participants were advised by a dietitian to reduce their daily caloric intake from sugars by 50% for 12 weeks.
  Interventions: Behavioral: 50% sugar reduction
- unmodified diet (No Intervention): Participants maintained an unmodified diet.

INTERVENTIONS:
Behavioral: 50% sugar reduction — Participants were advised by a dietitian to reduce their daily caloric intake from sugars by 50% for 12 weeks.
  Arms: 50% sugar reduction

SUMMARY:
The goal of this clinical trial is to determine whether reducing sugar intake by 50% for 12 weeks can change sweet taste perception in healthy adults and its consequences. The main questions it aims to answer are:

* Does sweet intensity change after reducing daily sugar intake by 50% for 12 weeks?
* How does sweet intensity change after completing dietary modification for 8 weeks?
* Does individual daily sugar intake change after completing dietary modification for 8 weeks?

Researchers will compare reducing daily sugar intake by 50% for 12 weeks to an unmodified diet to see if sugar reduction can change sweet intensity.

Participants will:

* Reduce daily sugar intake by 50% or maintain an unmodified diet for 12 weeks.
* Visit the clinic three times for anthropometric measurements, sweet perception tests, and to complete questionnaires.
* Keep a diet record for a total of 15 days during the research period.

ELIGIBILITY:
Inclusion Criteria:

* People with a fasting blood sugar level below 126 mg/dL or an HbA1C below 6.5% in the past 6 months, who are not currently being treated for diabetes.
* People who score 10 or more points on the sweet food consumption behavior questionnaire.
* People who are able to communicate in the Thai language.
* People who are able to chat and use video calls via the Line application.
* People who agree to modify their diet and beverages according to the recommendations of a dietitian.
* People who agree to undergo sweet taste testing, complete a food record, and fill out a questionnaire.

Exclusion Criteria:

* People with uncontrolled chronic conditions who have had changes in their treatment within the past 3 months.
* People with a history of severe illness in the past 6 months.
* People who regularly use medication, excluding contraceptives and vitamins.
* Pregnant women.
* People who have experienced a weight change of at least 10% over the past 3 months.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Sweet intensity change from baseline after 12 weeks of the intervention. | 16 weeks from baseline (12 weeks after the start of the intervention)
  Percentage of participants whose sweet intensity has increased after reducing daily sugar intake by 50% for 12 weeks, compared to those with an unmodified diet.

SECONDARY OUTCOMES:
Sweet intensity change from baseline after completing the intervention for 8 weeks. | 24 weeks from baseline
  Percentage of participants whose sweet intensity increased after completing dietary modification for 8 weeks, compared to those with an unmodified diet.
Changes in sugar consumption behavior from baseline | 24 weeks from baseline
  The average daily caloric intake from sugars after completing dietary modification for 8 weeks, compared to before the dietary change.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided